CLINICAL TRIAL: NCT07022379
Title: Real-word Assessment of the Clinical Characteristics and Adherence to the European Society of Cardiology Guideline-Directed Medical Therapies in Heart Failure Care Management in France: REMOTE-HF Study.
Brief Title: Adherence to European Society of Cardiology Guideline-directed Medical Therapies for Patients With Chronic Heart Failure in France
Acronym: GDMTs
Status: Completed | Type: Observational
Sponsor: Sophie NISSE-DURGEAT (Industry)
Responsible Party: Sponsor-Investigator, Sophie NISSE-DURGEAT, Nicolas Girerd, Satelia
Organization: Satelia (Industry)
Other Study IDs: 2024-REMOTE-HF
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Heart Failure With Preserved Ejection Fraction (HFPEF); Heart Failure With Reduced Ejection Fraction; Remote Monitoring; Care Management, Patient
Keywords: heart failure; guideline-directed medical therapy; GDMT; remote monitoring
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart failure patients remotely monitored with Satelia® Cardio program with SGLT2i treatment: Heart failure patients remotely monitored with Satelia® Cardio program without SGLT2i treatment

SUMMARY:
The goal of this observational study was to evaluate trends and determinants of SGLT2 inhibitor (SGLT2i) prescriptions in heart failure patients from 2021 to 2024, particularly in relation to LVEF subgroups and evolving scientific evidence (EMPEROR-Preserved, DELIVER, 2023 Guidelines).

Participant population were adults with heart failure using the Satelia®Cardio web application to remotely monitor their condition.

The main questions it aims to answer are:

* to compare the prescription of treatments (including doses, and distribution of patients according to various therapeutic classes recommend for heart failure) with ESC recommendations to see to what extent GDMTs are adhered to.
* to quantify the association between the presence of treatments and the risk of alerts/hospitalizations and overall death and as a function of LVEF using telemonitoring.
* to evaluate the adherence across patient profiles and cardiologist practices (outpatient vs. hospital-based).

Participants will complete follow-up, quality-of-life and patient support questionnaires and provide data regarding their treatments on the web application.

DETAILED DESCRIPTION:
A retrospective, multicenter descriptive study was conducted in France from January 1, 2021 to December 31, 2024. The REMOTE-HF study included 17,551 patients enrolled in remote monitoring program for heart failure (HF) management. We described and analyzed the implementation of ESC guidelines in patients monitored remotely with a web application named Satelia®Cardio (NP Medical).

Key clinical parameters such as age, gender, NYHA class, LVEF, and HF etiology were analyzed. Prescribed therapies including ACEi/ARB/ARNis, beta-blockers, MRAs, and SGLT2 inhibitors, were compared against the European Society of Cardiology (ESC) guideline-directed medical therapies (GDMTs).

Adherence was evaluated across patient profiles and cardiologist practices (outpatient vs. hospital-based) in France.

ELIGIBILITY:
Inclusion Criteria:

* registered to use Satelia®Cardio to remotely monitor their condition
* patients diagnosed with heart failure whatever the aetiology:

Especially patients who undergone:

Hospitalization within the previous 12 months, OR patients with NYHA class II or more, and BNP > 100 pg/ml OR NT-proBNP > 1000 pg/ml.

Exclusion Criteria:

* People aged under 18 years old
* Pregnant women
* Physical or psychological impossibility for the patient or carer to use the digital medical device according to the judgment of the doctor wishing to include the patient in the remote medical monitoring project.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with heart failure whatever the aetiology in France:
  Especially patients who undergone:
  Hospitalization within the previous 12 months, OR patients with NYHA class II or more, and BNP > 100 pg/ml OR NT-proBNP > 1000 pg/ml.Adult patients with heart failure in France.
Sampling Method: Probability Sample
Enrollment: 17551 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate trends and determinants of SGLT2 inhibitor (SGLT2i) prescriptions in heart failure patients. | From January 2021 to December 2024.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Affairs Department, NP Medical, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Girerd N, Barbet V, Seronde MF, Benchimol H, Jagu A, Tartiere JM, Hanon O, Picard F, Lafitte S, Lemaitre M, Pages N, Nisse-Durgeat S, Jourdain P. Association of a remote monitoring programme with all-cause mortality and hospitalizations in patients with heart failure: National-scale, real-world evidence from a 3-year propensity score analysis of the TELESAT-HF study. Eur J Heart Fail. 2025 Sep;27(9):1658-1669. doi: 10.1002/ejhf.3563. Epub 2025 Jan 14. PMID 39807086